CLINICAL TRIAL: NCT00001206
Title: Biological Markers in Childhood Psychiatric Disorders
Brief Title: Biological Markers in Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 850115; 85-M-0115
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2017-05-15

CONDITIONS: Attention Deficit and Disruptive Behavior Disorder; Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; Disruptive Behavior Disorders; Cerebrospinal Fluid; Lumbar Puncture; CSF; Longitudinal Prospective Follow-Up; Psychosocial Functioning; Risk Factors; Genetics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Attention Deficit and Disruptive Behavior Disorders

SUMMARY:
The purpose of this study is to evaluate individuals with Attention Deficit/Hyperactivity Disorder (ADHD) to learn more about the genetics of the disease.

This study is part of other ongoing studies of individuals with ADHD. The study participants have already undergone neurobiological measurements, particularly magnetic resonance imaging (MRI) of the brain, through other research studies. As a follow-up to these studies, participants will next undergo psychiatric interviews, neuropsychological tests, and another MRI. In addition to the clinical evaluation of the participants, further research will be conducted on the genetics of ADHD. These genetic studies will evaluate people with ADHD as well as their family members and a control group of healthy people.

DETAILED DESCRIPTION:
This protocol allows the continuing prospective longitudinal study of ADHD probands for whom we have neurobiological measures, particularly quantitative brain MRI. The follow-up consists of structured psychiatric interviews, and neuropsychological tests. Repeat MRI scans are obtained through protocol 89-M-0006.

The second purpose of this protocol is a study of the genetics of Attention-Deficit/Hyperactivity Disorder (ADHD). Subjects who have ADHD, their family members, and controls are studied under this protocol.

ELIGIBILITY:
* INCLUSION REQUIREMENTS-PROBANDS:

Current age of index probands: 15.21 plus or minus 3.42; previous participation in the NIMH Child Psychiatry Branch ADHD study.

Age adjusted dimensional ratings (Conners Rating Scales-Revised, and Strengths and Weaknesses of ADHD and Normal Behavior (SWAN)) of hyperactivity/impulsivity greater than or equal to 95th percentile for index and second sibling. Primary ratings for the index proband will be provided by main teacher.

Up to 150 ADHD probands for reassessment.

Consent and assent obtained in writing.

EXCLUSION CRITERIA - PROBANDS:

Presence of other known genetic conditions that are likely to be etiologic.

Onset of medical conditions that could produce symptoms of ADHD through non-genetic mechanisms (e.g., thyroid disorders, seizure disorders, inborn errors of metabolism, extremely low birth weight (less than 1000 gm), meningitis, intracranial pathology).

Presence of other psychiatric disorders that can produce symptoms similar to ADHD (e.g., major depression, bipolar disorder, severe anxiety disorders, pervasive developmental disorders, psychotic disorders, post-traumatic stress disorder).

Presence of neuropsychiatric conditions that may confound evaluation of ADHD (e.g., Tourette's syndrome, obsessive-compulsive disorder, or PANDAS (pediatric autoimmune neuropsychiatric disorders associated with streptococcus), intelligence quotient less than 80, reading achievement standard scores less than 75 or reading-intelligence discrepancy greater than 2 SD).

INCLUSION REQUIRMENTS-RELATIVES:

Subjects must be relatives of probands.

Consent and assent obtained in writing.

INCLUSION REQUIREMENTS -NORMAL VOLUNTEERS:

Up to 150 newly accrued normal volunteers unrelated to probands.

Same age range as probands.

Parent and teacher ratings within one SD of population means on ADHD/hyperactivity factors.

Consent and assent obtained in writing.

EXCLUSIONS - NORMAL VOLUNTEERS:

Presence of ADHD.

Presence of any other psychiatric disorders on structured psychiatric interview (DICA-IV).

Presence of known genetic conditions.

Onset, presence or history of medical conditions that could produce symptoms of ADHD through non-genetic mechanisms (e.g., thyroid disorders, seizure disorders, inborn errors of metabolism, extremely low birth weight (less than 1000 gm), meningitis, intracranial pathology).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 347 (Actual)
Dates: Start 1985-06-05; Study Completion 2017-05-15

CONTACTS AND LOCATIONS:
Overall Officials: Judith L Rapoport, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hauser ER, Boehnke M, Guo SW, Risch N. Affected-sib-pair interval mapping and exclusion for complex genetic traits: sampling considerations. Genet Epidemiol. 1996;13(2):117-37. doi: 10.1002/(SICI)1098-2272(1996)13:23.0.CO;2-5. PMID 8722742
- [Background] Thapar A, Hervas A, McGuffin P. Childhood hyperactivity scores are highly heritable and show sibling competition effects: twin study evidence. Behav Genet. 1995 Nov;25(6):537-44. doi: 10.1007/BF02327577. PMID 8540892
- [Background] LaHoste GJ, Swanson JM, Wigal SB, Glabe C, Wigal T, King N, Kennedy JL. Dopamine D4 receptor gene polymorphism is associated with attention deficit hyperactivity disorder. Mol Psychiatry. 1996 May;1(2):121-4. PMID 9118321